CLINICAL TRIAL: NCT01900808
Title: Improvement of Transient Elastography Applicability and Diagnostic Accuracy to Identify Significant Fibrosis by Experienced Operators Using the M and XL Probe.
Status: Completed | Type: Observational
Sponsor: Parc de Salut Mar (Other)
Responsible Party: Principal Investigator, José Antonio Carrion, MD, Parc de Salut Mar
Other Study IDs: APPLICABILITY- TE
Record Dates: First submitted 2013-07-12; First posted 2013-07-16 (Estimated); Last update posted 2016-01-18 (Estimated); Status verified 2013-07

CONDITIONS: Chronic Liver Diseases (CLD)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with chronic liver disease
  Interventions: Device: Trained operator with M probe.; Device: Experienced operator with M probe.; Device: Experienced operator with XL probe.

INTERVENTIONS:
Device: Trained operator with M probe. — Trained operator with M probe: non-drug intervention, baseline comparator.
Device: Experienced operator with M probe. — Experienced operator with M probe: non-drug intervention, longitudinal comparator.
Device: Experienced operator with XL probe. — Experienced operator with XL probe: non-drug intervention, longitudinal comparator.

SUMMARY:
Transient elastography (TE)is the reference method to identify liver stiffness (LSM) but fails to obtain a measurement in 3% of cases and results are considered unreliable in 16%. The aim of this study is to evaluate the applicability and diagnostic accuracy of TE performed by trained operators (<500 explorations), after a second evaluation by experienced explorers (>500 explorations) and after a third exploration using XL probe. Inadequate LSM will be re-evaluated by experienced operators with the M (standard size) probe. A third register will be performed with XL (obese size) probe in those patients with inadequate M probe determination. Diagnostic accuracy will be estimated in patients with liver biopsy to identify significant fibrosis with a TE cut-off value of 7.6 kPa (kilo pascal).

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic liver disease evaluated with TE by trained operators (experience <500 explorations).
* Signed inform consent.
* Aged between 18-90.

Exclusion Criteria:

* Patients with ascites.
* Pregnancy.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with liver stiffness
Sampling Method: Non-Probability Sample
Enrollment: 868 (Actual)
Dates: Start 2012-03; Primary Completion 2012-04 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Applicability of transient elastography (TE) | Will be calculated after evaluation of all included patients with M probe by trained operators (at baseline and after 48 weeks), M probe by experienced operators after 72 weeks and XL probe after 72 weeks.
  Applicability will be calculated as the proportion of reliable liver stiffness measurements (LSM). TE will be considered ADEQUATE when it included at least 10 valid measurements with a success rate ≥60% and interquartile range/median of LSM (IQR/M) ≤30% OR INADEQUATE.

SECONDARY OUTCOMES:
Diagnostic accuracy of TE | Will be calculated after evaluation of all included patients with M probe by trained operators after 48 weeks, M probe by experienced operators after 72 weeks and XL probe after 72 weeks.
  Diagnostic accuracy will be calculated with the number of correctly classified patients (wuth significant fibrosis) considering a cut-off value of 7.6 kPa.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital del Mar, Servei de Digestiu, Barcelona, Barcelona, Spain

REFERENCES:
- [Derived] Carrion JA, Puigvehi M, Coll S, Garcia-Retortillo M, Canete N, Fernandez R, Marquez C, Gimenez MD, Garcia M, Bory F, Sola R. Applicability and accuracy improvement of transient elastography using the M and XL probes by experienced operators. J Viral Hepat. 2015 Mar;22(3):297-306. doi: 10.1111/jvh.12296. Epub 2014 Aug 27. PMID 25164560